CLINICAL TRIAL: NCT02355366
Title: Family Focused Therapy (FFT) for Adolescents at Familial Risk for Bipolar
Brief Title: Family Focused Therapy for Teens at Risk for Bipolar Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Benjamin Goldstein, Associate Professor, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 404-2014
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Bipolar Disorder
Keywords: Offspring; significant mood symptoms
MeSH Terms: conditions — Bipolar Disorder | interventions — Family Therapy; Psychosocial Intervention; Psychotherapy; Behavior Therapy; Diagnostic Self Evaluation; Crew Resource Management, Healthcare

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Focused Therapy (FFT) (Experimental): Participants will receive Family-Focused Therapy (FFT). It will consist of twelve, 1-hour long sessions, over a period of 4 months. The 12 sessions will include psychoeducation (sessions 1-4), training in communication enhancement (sessions 5-8) and training in relation to problem-solving skills (sessions 9-12).
  Interventions: Behavioral: Family-Focused Therapy
- Brief Educational Treatment (Active Comparator): Participants will be receive 1-2 educational sessions which will include diagnostic feedback, recommendations for further treatment and crisis intervention if required.
  Interventions: Behavioral: Brief Educational Treatment

INTERVENTIONS:
Behavioral: Family-Focused Therapy — Family Focused Therapy is a manual-based, psycho-educational intervention which is designed to reduce intra-familial stress, conflict, and affective arousal by enhancing communication and problem solving skills among families who are affected by bipolar disorder (Miklowitz et al., 2013). It concentrates on skills relevant to managing the prodromal stages of bipolar disorder, such as mood monitoring, reducing family conflict, improving problem solving, stabilizing daily routines and regulating sleep/wake cycles (Miklowitz, 2012).
  Other Names: FFT; Family Therapy; Psychosocial Intervention; Psychoeducaton; Psychotherapy; Behaviour Therapy
  Arms: Family Focused Therapy (FFT)
Behavioral: Brief Educational Treatment — Brief Educational Treatment will consist of 1 - 2 sessions involving both parents and adolescents; it will consist of diagnostic feedback following the adolescent's baseline assessment. It will provide families with information and strategies on tracking and managing adolescent mood disorders. Additionally, ongoing medication management and crisis family sessions will be available if required.
  Other Names: Psychoeducation; Diagnostic Evaluation; Crisis Management
  Arms: Brief Educational Treatment

SUMMARY:
The present study aims to examine the effects of a 4 month, family focused therapy (FFT) intervention on the 1 year course of mood symptoms in offspring of parents with bipolar disorder (BD). The study will also examine the level of expressed emotion among families and how this impacts on FFT treatment outcomes. This study seeks to replicate a previous study by Miklowitz, Schneck, Singh, Taylor, George and colleagues (2013), which demonstrated the efficacy of FFT among BD offspring. Importantly, the present study will introduce biological measures that predict and reflect improvement in symptoms and expressed emotion. These markers reflect stress-related biological systems and include saliva samples to ascertain cortisol, interleukin-6 (IL-6) and salivary alpha amylase (sAA).

DETAILED DESCRIPTION:
Children of parents with bipolar disorder (BD) have increased risk of developing BD themselves. BD in youth is associated with increased risk for suicidality, psychosis, substance abuse and compromised psychosocial functioning. In addition, offspring of parents with BD have an increased vulnerability for developing other psychopathology (e.g. major depression). At present, research examining early intervention and treatment for this high risk population is limited. However, a recent study in symptomatic youth at risk for BD indicated that participation in a family focused therapy (FFT) intervention led to positive treatment outcomes. The present study aims to examine the effects of FFT in BD offspring in comparison to a brief educational treatment. Specifically, this study will examine whether FFT can have protective effects on individuals' mood symptoms and functioning by targeting the family environment. We will expand upon previous research by also measuring biological markers of stress (i.e., cortisol levels) and changes in family functioning over time. With this knowledge, the results of this study may help to shed light on the importance of early intervention and improve preventative treatment options for youth at high-risk for bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking males and females of any race/ethnicity
2. 13-19 years of age
3. Have at least 1 biological parent who meets diagnostic criteria for bipolar disorder (BD) type I or II, based on the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I)
4. Adolescent is experiencing current, significant mood symptoms indicated by a psychiatric status rating (PSR) score of 3
5. At least 1 parent/primary caregiver is available to attend sessions.

All participants will complete rigorous diagnostic interviews to ensure that they meet these requirements.

Exclusion Criteria:

1. Unable to provide informed consent (e.g., severe psychosis, developmental delay)
2. Have met the DSM-IV criteria (based on the Schedule for Affective Disorders and Schizophrenia for School Age Children, Present and Life Version - K-SADS-PL), for substance dependence in the past 3 months (excluding nicotine dependence)
3. Are victims of current sexual or physical abuse by parents or live among domestic violence
4. For offspring, already meet criteria for bipolar disorder (BD) type I or II.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04; Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
KSADS Mania Rating Scale (KMRS) | Change from baseline to endpoint (assessed at 0, 4, 8 and 12 months)
  Measures symptom severity.
KSADS Depression Section (KDRS) | Change from baseline to endpoint (assessed at 0, 4, 8 and 12 months)
  Measures symptom severity.
Adolescent Longitudinal Interval Follow-up Evaluation (A-LIFE) | Change from baseline to endpoint (assessed at 0, 4, 8 and 12 months)
  Used to track symptom severity, treatment (both psychosocial and psychotropic), self-injurious/suicidal behavior and psychosocial functioning over time.
The Family Environment Scale (FES) | Change from baseline to endpoint (assessed at 0, 4, 8 and 12 months)
  Examines each family member's perceptions of the family in three ways-as it is (real), as it would be in a perfect situation (ideal) and as it will probably be in new situations (expected).
Family Adaptability & Cohesion & Adaptability Scale (FACES) | Change from baseline to endpoint (assessed at 0, 4, 8 and 12 months)
  Evaluate the adaptability and cohesion dimensions in family interactions.
Conflict Behaviour Questionnaire (CBQ) | Change from baseline to endpoint (assessed at 0, 4, 8 and 12 months)
  Measures conflict and negative communication between parents and adolescents.
Issues Checklist | Change from baseline to endpoint (assessed at 0, 4 and 12 months)
  Measures potential areas of conflict between parents and adolescents.
Cortisol | Change from baseline to endpoint (assessed at 0, 4, and 12 months)
  Stress-related biomarker obtained through saliva samples.
Interleukin 6 (IL-6) | Change from baseline to endpoint (assessed at weeks 0, 4, and 12 months)
  Stress-related biomarker obtained through saliva samples.
Alpha Amylase | Change from baseline to endpoint (assessed at 0, 4, and 12 months)
  Stress-related biomarker obtained through saliva samples.
Five Minute Speech Sample | Change from baseline to endpoint (assessed at 0, 4, and 12 months)
  Assesses level of expressed emotion (EE) within the parental household.
Emotional Response to Conflict Scale (ERCS) | Change from baseline to endpoint (assessed at 0, 4 and 12 months)
  Assesses individuals' emotional responses to a brief, laboratory based, conflict negotiation task.

SECONDARY OUTCOMES:
Children Global Assessment Scale | Change from baseline to endpoint (assessed at 0, 4, 8 and 12 months)
  Quantifies overall level of functioning for a child or adolescent during a specified time period.
Anthromorphic Data | Change from baseline to endpoint (Assessed at weeks 0 and 12 months)
  Measures height, weight, body mass index, & blood pressure.
Working Alliance Inventory Short-Revised (WAI-SR) | Change from baseline to endpoint. For FFT Group: Assessed after therapy sessions 1, 4, 8 & 12. For Education Control Group: Assessed after therapy sessions 1 & 2.
  Measures therapeutic alliance.
General Information Sheet | Baseline
  Demographics

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Goldstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Miklowitz DJ, Schneck CD, Singh MK, Taylor DO, George EL, Cosgrove VE, Howe ME, Dickinson LM, Garber J, Chang KD. Early intervention for symptomatic youth at risk for bipolar disorder: a randomized trial of family-focused therapy. J Am Acad Child Adolesc Psychiatry. 2013 Feb;52(2):121-31. doi: 10.1016/j.jaac.2012.10.007. Epub 2013 Jan 2. PMID 23357439
- [Background] Miklowitz DJ. Family-focused treatment for children and adolescents with bipolar disorder. Isr J Psychiatry Relat Sci. 2012;49(2):95-101. PMID 22801288